CLINICAL TRIAL: NCT07044115
Title: A Phase 1b/2 Clinical Study Evaluating the Tolerance, Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of Recombinant Humanized Monoclonal Antibody MIL62 Injection in Subjects With Lupus Nephritis
Brief Title: Evaluation of the Tolerance, Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of MIL62 Injection for Treating Lupus Nephritis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MIL62-CT203
Record Dates: First submitted 2025-06-23; First posted 2025-06-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis; CD20 monoclonal antibody; MIL62
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIL62 (Experimental)
  Interventions: Drug: Recombinant Humanized Monoclonal Antibody MIL62 Injection
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Recombinant Humanized Monoclonal Antibody MIL62 Injection — Phase 1b:
  Intravenous infusion. Dose group 1 (500mg), dose group 2 (1000mg); administered on Day 1 of Weeks 1, 3, 25, 27, 53, 55, and 77. Dose group 3 (500mg), administered on Days 1, 2, 3, 4, 25, 26, 27, 28, 53, 54, 55, 56, 77, and 78 of each respective week.
  Phase 2:
  Use the dose and frequency determined in Phase 1b.
  Arms: MIL62
Drug: placebo — Phase 1b:
  Intravenous infusion. Dose group 1 (500mg), dose group 2 (1000mg); administered on Day 1 of Weeks 1, 3, 25, 27, 53, 55, and 77. Dose group 3 (500mg), administered on Days 1, 2, 3, 4, 25, 26, 27, 28, 53, 54, 55, 56, 77, and 78 of each respective week.
  Phase 2:
  Use the dose and frequency determined in Phase 1b.
  Arms: placebo

SUMMARY:
This study is composed of two stages: Part A is a randomized, double-blind, placebo-controlled dose-escalation study (i.e., Phase 1b study). The first part has a total of 3 dose groups, with 10 subjects enrolled in each dose group. Subjects are randomly assigned to receive MIL62 combined with standard of care or placebo combined with standard of care at a 4:1 ratio. Based on the tolerability, safety, pharmacodynamics, pharmacokinetics, and preliminary efficacy of the 3 dose groups, the maximum tolerated dose (MTD), recommended phase 2 dose (RP2D), and dosing frequency will be determined.

Part B is open-label, enrolling 10 subjects who will receive the recommended dose of MIL62 combined with standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and <75 years, gender not restricted;
2. Diagnosed with systemic lupus erythematosus (SLE) according to the 2019 European League Against Rheumatism (EULAR) / American College of Rheumatology (ACR) classification criteria;
3. Urinary protein/creatinine ratio (UPCR) > 1.0 (24-hour urine);
4. If the patient is taking drugs that may affect kidney function (e.g., ACE inhibitors, cholesterol-lowering drugs), the dosage must remain stable for at least 4 weeks prior to enrollment and throughout the study;
5. No need to receive vaccination during the study or need vaccination only after at least 16 weeks following the last dose of study drug;
6. Signed written informed consent.

Exclusion Criteria:

1. Screening reveals other severe kidney diseases or conditions, including: ① Need for dialysis or transplant therapy; ② Kidney biopsy within the last 6 months shows more than 50% glomerulosclerosis;
2. Screening reveals the following diseases or conditions: ① Other autoimmune diseases besides SLE; ② Clinically significant bleeding risks, or conditions requiring plasma exchange, blood transfusion, or platelet transfusion;
3. Positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb), with HBV DNA levels outside normal range; positive for HCV antibody and HCV RNA; positive for HIV serum reaction; positive for syphilis test;
4. Pregnant and breastfeeding women; for women of childbearing potential who have not undergone sterilization: unwilling to use appropriate contraception methods (e.g., oral contraceptives, intrauterine devices, or barrier methods with spermicide) during the treatment period and for at least 18 months after the last dose of study drug;
5. For men who have not undergone sterilization: unwilling to use barrier contraception during the study and for at least 18 months after the last dose of study drug, and unwilling to have their spouse use other contraception methods;
6. The investigator considers other situations not suitable for participation in the study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects achieving complete renal remission (CRR) at 76 weeks | week 76
  Percentage of Participants with UPCR < 0.3 and estimated glomerular filtration rate (eGFR) decline ≤ 15% from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China